CLINICAL TRIAL: NCT06968910
Title: Cannabidiol-based Therapy to Attenuate Non-bacterial Prostatitis Symptoms - Single-arm Open-label Pilot Clinical Trial With Intrarectal Administration
Brief Title: CBD-based Therapy to Attenuate Non-bacterial Prostatitis Symptoms
Acronym: Urol-CBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palacky University (Other)
Collaborators: CB21 Pharma Ltd. (Unknown)
Responsible Party: Principal Investigator, Jan Vacek, Olomouc University Hospital, Palacky University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 176/22
Record Dates: First submitted 2025-04-26; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Prostatitis
Keywords: prostatitis; chronic pelvic pain; cannabidiol and hyaluronic acid; rectal delivery
MeSH Terms: conditions — Prostatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CBD-based therapy (Experimental): Participants self-administered nightly intrarectal cannabidiol (CBD)-based suppositories for 30 consecutive days.
  Interventions: Device: CANNEFF® SUP rectal suppositories

INTERVENTIONS:
Device: CANNEFF® SUP rectal suppositories — CANNEFF® SUP suppositories with cannabidiol (CBD = 100 mg) and hyaluronic acid (HA = 6.6 mg) as active ingredients

SUMMARY:
Efficacy and safety of the medical device rectal CANNEFF® SUP suppositories containing two active ingredients cannabidiol (CBD) and hyaluronic acid (HA) in alleviating non-bacterial prostatitis symptoms and improving quality of life in men will be evaluated.

DETAILED DESCRIPTION:
Chronic non-bacterial prostatitis/chronic pelvic pain syndrome (CP/CPPS) is the third most common urogenital diagnosis in men, following benign prostatic hyperplasia and prostate cancer, with an estimated prevalence reaching 8.2%. Clinically, CP/CPPS often presents with persistent pelvic pain, lower urinary tract symptoms (LUTS), and sexual dysfunction, all of which can substantially diminish quality of life. Psychological comorbidities, including anxiety, stress, and depression, further amplify the burden on patients. Despite its considerable socioeconomic impact, no definitive treatment consensus exists for CP/CPPS. This study assessed the effects of rectal administration of cannabidiol (CBD)-based therapy in men with CP/CPPS. A single-arm, open-label pilot trial on men with CP/CPPS (NIH Chronic Prostatitis Symptom Index [NIH-CPSI] >10, pain subscore ≥4). The participants self-administered rectal CANNEFF® suppositories containing CBD (100 mg) and hyaluronic acid (HA = 6.6 mg) as active ingredients, nightly for 30 days. Outcome measures included changes in NIH-CPSI total score, International Prostate Symptom Score (IPSS), and International Index of Erectile Function (IIEF-5). Safety and tolerability were assessed.

ELIGIBILITY:
Inclusion Criteria:

* men aged 18-50 years
* reported pelvic pain for ≥3 months in the past 6 months
* reported the National Institutes of Health Chronic Prostatitis Symptom Index (NIH-CPSI) total score >10 with a pain subscore ≥4
* clinically and laboratory diagnosed CP/CPPS

Exclusion Criteria:

* confirmed genitourinary infections (e.g., Escherichia coli, Enterococcus faecalis, Chlamydia spp.)
* recent antibiotic use (within 6 months)
* cannabis use
* alpha-blockers or phytotherapeutics in the preceding 4 weeks
* no history of pelvic trauma, surgery or radiotherapy, neurogenic bladder, post-void residual >50 mL, or psychiatric disorders affecting compliance

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only biological male identity.
Enrollment: 35 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Alleviating Chronic Non-bacterial Prostatitis Symptoms | 30 days
  The primary outcome was the change in NIH Chronic Prostatitis Symptom Index (NIH-CPSI) total score between baseline (Day 0) and Day 30. The NIH-CPSI has a total score range from 0 to 43, and it includes three subscales addressing pain (score range 0-21), urinary symptoms (score range 0-10), and quality of life (QOL) (score range 0-12). Higher score means a worse outcome.
Alleviating Chronic Pelvic Pain Symptoms | 30 days
  The changes in the NIH-CPSI pain subscore (score range 0-21) were evaluated to capture the specific impact on pelvic pain. Higher score means a worse outcome.

SECONDARY OUTCOMES:
International Prostate Symptom Score Evaluation | 30 days
  Secondary outcome measures included the International Prostate Symptom Score (IPSS). The IPSS evaluates lower urinary tract symptoms (both storage and voiding). A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms. The index was assessed at baseline and again on Day 30.
Erectile Function Evaluation | 30 days
  The five-item International Index of Erectile Function (IIEF-5) was evaluated, whereas the IIEF-5 provides a brief assessment of erectile function (higher scores indicating better function). Interpretation: score 22-25 - No erectile dysfunction, 17-21 - Mild erectile dysfunction, 12-16 - Mild to moderate erectile dysfunction, 8-11 - Moderate erectile, 5-7 - Severe erectile dysfunction. The index was assessed at baseline and again on Day 30.
Safety Profile Evaluation | 30 days
  Adverse events reported were monitored after 30 d of intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, University Hospital Olomouc, Czech Republic, Olomouc, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosen RC, Riley A, Wagner G, Osterloh IH, Kirkpatrick J, Mishra A. The international index of erectile function (IIEF): a multidimensional scale for assessment of erectile dysfunction. Urology. 1997 Jun;49(6):822-30. doi: 10.1016/s0090-4295(97)00238-0. PMID 9187685
- [Background] Barry MJ, Fowler FJ Jr, O'Leary MP, Bruskewitz RC, Holtgrewe HL, Mebust WK, Cockett AT. The American Urological Association symptom index for benign prostatic hyperplasia. The Measurement Committee of the American Urological Association. J Urol. 1992 Nov;148(5):1549-57; discussion 1564. doi: 10.1016/s0022-5347(17)36966-5. PMID 1279218
- [Background] Litwin MS, McNaughton-Collins M, Fowler FJ Jr, Nickel JC, Calhoun EA, Pontari MA, Alexander RB, Farrar JT, O'Leary MP. The National Institutes of Health chronic prostatitis symptom index: development and validation of a new outcome measure. Chronic Prostatitis Collaborative Research Network. J Urol. 1999 Aug;162(2):369-75. doi: 10.1016/s0022-5347(05)68562-x. PMID 10411041
- [Background] Nickel JC, Downey J, Hunter D, Clark J. Prevalence of prostatitis-like symptoms in a population based study using the National Institutes of Health chronic prostatitis symptom index. J Urol. 2001 Mar;165(3):842-5. PMID 11176483